CLINICAL TRIAL: NCT04770181
Title: Effects of Cranial Electrotherapy Stimulation on Psychological Distress and Maternal Functioning in New Mothers During the Postpartum Period
Brief Title: New Mothers Alpha-Stim
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled and will not be restarted.
Sponsor: Christina Murphey, RN, PhD (Individual)
Responsible Party: Sponsor-Investigator, Christina Murphey, RN, PhD, Associate Professor, Murphey, Christina, RN, PhD
Organization: Murphey, Christina, RN, PhD (Individual)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCHIRB#00001244
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-11

CONDITIONS: Anxiety; Depression; Insomnia; Sleep Quality
Keywords: Cranial Electrotherapy Stimulation (CES); Efficacy; Post Partum; Anxiety; Depression; Insomnia; Sleep Quality; Maternal Functioning
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The design for the proposed study is a matched-pair, quasi-experimental, 1:1 randomized, double-blind, sham-controlled clinical trial with a longitudinal component. The analytic technique employed to answer the research questions will be repeated measures analysis of covariance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blocked randomization method will be used to assign participants to active and sham groups. Participants will be assigned to CES treatment or sham CES using a 1:1 ratio. Electromedical Products International, Inc. (EPI) will randomize the assignment of appropriate devices to active or sham groups by using a random list of computer generated numbers (1 for active and 2 for sham) in randomly selected block sizes. The PI and participants are blinded to which participants have Alpha-Stim® CES active or sham devices until data analysis is complete. After the completion of data analysis, blinding will be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Comparator (Active Comparator): About the size of a smart phone, the Alpha-Stim® AID CES device delivers a mild electrical current (100-500 µA) to the brain via ear clips electrodes. The active intervention is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks at 0.5 Hz. 50% duty cycle with a fixed current of 100 µA (subsensory level).
  Interventions: Device: Alpha-Stim AID CES (Active Comparator)
- Sham Comparator (Sham Comparator): The Alpha-Stim® AID CES sham device is identical in appearance to the active device but is inactive and does not emit electrical current to the brain via ear clip electrodes. The sham intervention is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks.
  Interventions: Device: Alpha-Stim AID CES (Sham Comparator)

INTERVENTIONS:
Device: Alpha-Stim AID CES (Active Comparator) — The Alpha-Stim® AID CES device delivers a mild electrical current (100-500 µA) to the brain via ear clips electrodes. The treatment regimen is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks at 0.5 Hz. 50% duty cycle with a fixed current of 100 µA (subsensory level).
  Other Names: Alpha-Stim AID
  Arms: Active Comparator
Device: Alpha-Stim AID CES (Sham Comparator) — The Alpha-Stim® AID CES sham device is inactive and does not emit electrical current to the brain via ear clip electrodes. The sham treatment regimen is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks.
  Other Names: Alpha-Stim AID
  Arms: Sham Comparator

SUMMARY:
The birth of a child is a major life event that can be filled with excitement, anticipation and joy. However, the transition and adaptation to new demands, roles, responsibilities, and changes in relationships can be stressful, especially for new mothers. In addition, new mothers typically encounter physiological changes and struggle with concerns about weight gain, body image, sexuality, and other physical difficulties such as fatigue. These problems may generate or exacerbate stress, lead to an actual or perceived crisis and psychological distress.

Psychological distress, defined as anxiety, depression, and insomnia, in this study, often increases during the postpartum period and can negatively affect maternal mental health status, maternal and family relationships, and infant-child health. The purpose of this study is to evaluate the effects of cranial electrotherapy stimulation (CES) on anxiety, insomnia, depression, and maternal functioning in first time new mothers following childbirth.

DETAILED DESCRIPTION:
The birth of a child is a major life event that can be filled with excitement, anticipation and joy. However, the transition and adaptation to new demands, roles, responsibilities, and changes in relationships can be stressful, especially for first-time mothers. In addition, new mothers typically encounter physiological changes and struggle with concerns about weight gain, body image, sexuality, and other physical difficulties such as fatigue. These problems may generate or exacerbate stress, lead to an actual or perceived crisis and psychological distress.

Psychological distress, defined as depression, anxiety and insomnia, in this study, often increases during the postpartum period and can negatively affect maternal mental health status, maternal and family functioning, and infant-child outcomes. These conditions commonly present as co-morbidities, but are often unrecognized in clinical practice or under-treated as co-morbidities in new mothers. This unrecognized cluster of co-morbidities may lead to psychological distress and subsequently poor outcomes for mothers, their infants and children.

Current treatment recommendations for depression, anxiety and insomnia are primarily pharmaceutical or psychotherapy, both of which have limitations related to cost, time involved and ineffectiveness for some women. Consequently, there is a need to examine other treatment approaches including complementary modalities, such as cranial electrotherapy stimulation (CES), particularly in light of current evidence that shows the efficacy of early detection, intervention and treatment for pregnant and postpartum women.

The primary objective of this study is to investigate the effect of CES on anxiety in new mothers following childbirth. The secondary objectives are to: (1) determine the effects of CES on depression and insomnia; (2) explore the effect of CES on maternal functioning in new mothers following childbirth, and (3) to examine if items 1 & 2 on the 14 item Hamilton Anxiety Rating Scale (HAM-A14) perform well as a screening test for anxiety. Please see the enclosed Instrument Description document for detailed information related to this scale.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a total score of ≥ 16 on the HAM-A14 and ≥2 on both Hamilton Anxiety Rating Scale (HAM-A14) item 1 (anxious mood) and item 2 (tension) at screening and baseline to be considered for inclusion into the study.
2. Participant is a primiparous new mother, 18-45 years inclusive, who had an uncomplicated vaginal or cesarean birth, gave birth to a healthy baby and both mother and baby are healthy at enrollment and randomization in the study.
3. Sexually active female participants of childbearing potential must be self-report practicing, at least, one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female participants of childbearing potential must have a negative urine pregnancy test before receiving study treatment.
4. Written informed consent must be obtained from the participant before study participation.
5. Participant is in good medical health.
6. No current abuse of alcohol or other substance.
7. Capable of giving informed consent.
8. Capable of doing active or sham CES treatments and completing all study requirements independently
9. For compliance, participants need to have completed 85% (36) of treatments to continue participation in the study

Exclusion Criteria:

1. Participant had serious complications during or after a vaginal or cesarean delivery.
2. Participant had multiple births.
3. Participant meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-V criteria for a mental disorder diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by medical history and/or self-report.
4. Participant is clinically judged by the investigator to be at risk for suicide or is acutely suicidal. Participant has attempted suicide one or more times within the past twelve months.
5. Participant has a Hamilton Anxiety Rating Scale (HAM-A14) score above 30 which suggests a very severe clinical level of anxiety symptoms.
6. Participant has a Hamilton Depression Rating Scale (HAM-D17) score above 30 which suggests a very severe clinical level of depressive symptoms.
7. Participant has a psychiatric condition that would require inpatient or partial psychiatric hospitalization.
8. Participant has a significant history of medical disease (i.e. cardiovascular, hepatic (e.g., cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological (seizures), gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
9. Participant is pregnant, planning to become pregnant. If a participant becomes pregnant, she will be dropped from the study immediately and followed appropriately.
10. Participant has had concomitant therapy with another investigational drug, or participation in an investigational drug study within one month before entering this study.
11. Participant has a history of poor compliance or in the investigator's judgment any participant who is not compliant with the requirements of the study.
12. Participant has had previous trial of CES.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To measure the effect of CES on anxiety in new mothers during the postpartum period. | Duration is six weeks
  The Hamilton Anxiety Rating Scale (HAM-A14)

SECONDARY OUTCOMES:
To measure the effect of CES on depression in new mothers during the postpartum period. | Duration is six weeks
  The Hamilton Depression Rating Scale17 (HAM-D17)
To measure the effect of CES on sleep quality in new mothers during the postpartum period. | Duration is six weeks
  The Pittsburgh Sleep Quality Index (PSQI19)
To measure the effect of CES on insomnia in new mothers during the postpartum period. | Duration is six weeks
  The Insomnia Severity Index (ISI7)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Murphey, RN, PhD, Principal Investigator — Texas A&M University - Corpus Christi
Locations (2):
- United States (2):
  - Primay care; OB-GYN Clinic, Austin, Texas
  - Primary care; OB-GYN Clinic, Corpus Christi, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphey C, Carter P, Price LR, Champion JD, Nichols F. Psychological Distress in Healthy Low-Risk First-Time Mothers during the Postpartum Period: An Exploratory Study. Nurs Res Pract. 2017;2017:8415083. doi: 10.1155/2017/8415083. Epub 2017 Jan 16. PMID 28191350